CLINICAL TRIAL: NCT06341868
Title: Dynamic Gait-Synchronous Neuromuscular Electrical Stimulation Following Anterior Cruciate Ligament Reconstruction
Brief Title: Dynamic Muscular Electrical Stimulation Following Anterior Cruciate Ligament Reconstruction in Military Academy Cadets
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Collaborators: Medical Technology Enterprise Consortium (Unknown)
Responsible Party: Principal Investigator, Shawn Gee, MD, MD, Keller Army Community Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KACH.2023.0067; 23KACH008 (Other: Keller Army Community Hospital)
Record Dates: First submitted 2024-03-18; First posted 2024-04-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: knee; Anterior Cruciate Ligament; Gait; Neuromuscular electric stimulation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care + KneeStim controlled low intensity (Sham Comparator): Low intensity range
  Interventions: Device: KneeStim
- Standard of Care + KneeStim flexible intensity (Experimental): Flexible to high intensity range
  Interventions: Device: KneeStim

INTERVENTIONS:
Device: KneeStim — Participant will be randomized to either be in control or experimental group

SUMMARY:
The goal of this clinical trial is to examine the effects of 12 weeks of post-operative use of a novel wearable electrical stimulation knee sleeve device (KneeStim) on post-operative biomechanical function (gait). Participants will be United States Military Academy cadets aged 17-27 years. The main questions it aims to answer are:

* Examine the effects of KneeStim wear on cadets' post-operative gait
* Examine changes in site-specific skeletal muscle mass
* Examine the changes in patient-reported outcomes
* Assess time to return to full duty
* Compare Bioelectrical Impedance Analysis (BIA) measurements to Magnetic Resonance Imaging (MRI) measurements (total thigh volume)
* Determine the concurrent criterion validity of the KneeStim device compared to gold- standard metrics (3D Motion Capture)

Participants will undergo body composition analysis, MRI, strength testing, standard of care rehabilitation, gait analysis, and complete surveys. Participants will wear the KneeStim during their standard of care rehabilitation visits for the first 5 weeks post-operative, and throughout daily tasks from 6-12 weeks.

Researchers will compare a control group (standard of care + KneeStim controlled low intensity) to an experimental group (standard of care + KneeStim flexible intensity) to assess the aims previously mentioned..

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) tears have a recovery time of nearly 6-12 months with operative treatment. While most service members return to full duty after ACL reconstruction, it is delayed by quadriceps activation, muscle weakness, and abnormal gait patterns. Neuromuscular electric stimulation devices are already being used in physical therapy to complement gains in muscle strength and size. The innovation of KneeStim, is that it can be used to stimulate knee muscles while the individual is engaging in their daily activities. This study looks at the effects of 12 weeks of post-operative use of the KneeStim on biomechanical function (gait) in United States Military Academy Cadets aged 17-27 years of age. The investigators hypothesize that using the KneeStim will accelerate normalization of the biomechanical function parameters of gait and thus return to full duty.

ELIGIBILITY:
Inclusion Criteria:

1. United States Military Academy cadet between ages of 17-27 years
2. Undergoing a Primary ACL Reconstruction, or Revision ACL Reconstruction

Exclusion Criteria:

1. Concomitant or prior high tibial osteotomy (HTO)
2. Concomitant or prior cartilage restoration procedure
3. Concomitant ligamentous reconstruction (lateral collateral ligament; posterior cruciate ligament; medial collateral ligament)
4. Contraindications to using the KneeStim device

   - Use of pacemaker, defibrillators, or other implanted electronic devices, as this may cause electric shock, burns, electrical interference, or death Unstable angina or decompensated heart failure Epilepsy or history of seizure disorder Pregnancy or planning to become pregnant (Self reported) Critical ischemia of lower limbs Moderate to severe dementia Altered sensation at the knee such that the user cannot feel a pinprick Undiagnosed pain syndromes
5. Any meniscus tear precluding weight bearing for 6 weeks.

Ages: 17 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in gait post-operatively assessed by the KneeStimTM Device | 6 weeks;3, 6, 9, 12 months post-operative
  Effects of a novel wearable electrical stimulation knee sleeve device (KneeStim) on post-operative biomechanical function (femur sagittal angle, tibial sagittal angle, femur coronal angle, tibial coronal angle, femur and tibia coronal velocity)

SECONDARY OUTCOMES:
change in gait post-operatively assessed by 3D Motion capture | 3, 6, 9, 12 months post-operative
  Kinetic and kinematic biomechanical data will be monitored throughout the return to run phases of rehabilitation in knee and hip joints (walking and running); changes in gait speed (walking and running); changes in join angle range of motion (walking and running); changes in stride length (walking and running)
change in gait post-operatively assessed by force plate instrumented treadmill | 3, 6, 9, 12 months post-operative
  Ground reaction forces will be recorded simultaneously with the motion capture system via force plates on an instrumented treadmill to determine force output between limbs during walking and running trials.
change in muscle volume assessed by MRI | pre-operative, 3, 6, 9, 12 months post-operative
  Summation of the cross-sectional area and volumetric measurements
ACL graft healing assessed by MRI | pre-operative, 3, 6, 9, 12 months post-operative
  Signal intensity will be used to monitor tissue quality throughout healing process
Change in isometric muscle strength assessed by CSMi HUMAC NORM | 3, 6, 9, 12 months post-operative
  Rate of torque development (in ms) over time.
Change in skeletal muscle mass assessed by bioelectrical impedance analysis (SECA BIA) | pre-operative, 4, 8 weeks; 3, 6, 9, 12 months post-operative
  Skeletal muscle mass will be measured (in kg) to monitor rate of muscle hypertrophy/atrophy over rehabilitation timeline.
Change in lean body mass assessed by bioelectrical impedance analysis (SECA BIA) | pre-operative, 4, 8 weeks; 3, 6, 9, 12 months post-operative
  Muscle mass, bone mass, and body fluid (kg/m2) will be measured to contribute to Body Mass Index (BMI) scores.
Change in fat mass assessed by bioelectrical impedance analysis (SECA BIA) | pre-operative, 4, 8 weeks; 3, 6, 9, 12 months post-operative
  Fat mass (kg/m2) will be measured to contribute to body mass index (BMI) scores.
Change in knee pain and function assessed by the Knee Injury and Osteoarthritis Score (KOOS) | pre-operative, 3, 6, 9, 12 months post-operative
  The KOOS is a self-reported outcome measure assessing the patient's perspective about the health, symptoms, and functionality of their knee. It is a 42-item questionnaire, including 5 subscales: symptoms, pain, activities of daily living, function in sports/recreation, and quality of life. A likert scale is used and all items have five possible answers ranging from 0 (no problems) to 4 (extreme problems). The five subscale scores are calculated as the sum of the items for each subscale. Scores are then transformed to a 0-100 scale, with 0 representing extreme knee problems and 100 representing no knee problems.
Change in knee pain and function assessed by the International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC) | pre-operative, 3, 6, 9, 12 months post-operative
  The IKDC is a self-reported outcome measure that assesses knee disability and function before and after treatment. It consists of 18 items that measure symptoms, function, and sports activity. Response types include 5-point Likert Scales, 11-point Likert scales, and dichotomous "yes-no" responses.
Change in knee pain assessed by the Patient-Reported Outcome Measure Information System (PROMIS-29) | pre-operative, 3, 6, 9, 12 months post-operative
  PROMIS-29 is a self-reported outcome measure assessing for the patient's pain intensity. It is a 28-item questionnaire, which includes 7 subscales of four items each: physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. A likert scale is used for all domain response scales, however they vary in responses.
Change in knee function assessed with the Single Assessment Numeric Evaluation Method (SANE) | pre-operative, 3, 6, 9, 12 months post-operative
  Participants will provide a numerical rating from 0 (least normal) to 100 (most normal) of the perceived improvement in knee health in relation to their pre-injury baseline.
Change in knee function assessed by the Marx Activity Rating Scale (MARS) | pre-operative, 3, 6, 9, 12 months post-operative
  MARS includes 4 items that assess the frequency of running, cutting, decelerating, and pivoting based on the subjects "healthiest and most active state in the past year". Each item is scored on a 5-point ordinal scale ranging from 0 (less than 1 time in a month) to 4 (4 or more times in a week), and the total scale score is obtained by summing the individual items' scores (range, 0-16). A higher score indicates more functional demand on the knee joint and potentially a higher risk of injury.
Impact of ACL surgery on overall quality of life assessed by the Anterior Cruciate Ligament-Quality of Life (ACL-QOL) | pre-operative, 3, 6, 9, 12 months post-operative
  The questionnaire consists of 32 equally weighted questions that are answered using a 100 mm visual analog scale and is scored of 100. It comprises 5 domains, including (1) symptoms and physical complaints (5 items); (2) work-related concerns (4 items); (3) recreational activity and sport participation or competition (12 items); (4) lifestyle (6 items); and (5) social and emotional (5 items).
Change of running gait function from the patients' perspective assessed by the University of Wisconsin Running Injury and Recovery Index (UWRI) | pre-operative, 3, 6, 9, 12 months post-operative
  The 9-item UWRI assesses running ability following a running related injury, with the maximum score of 36 indicating a return to preinjury running ability.
Change of knee pain from the patients' perspective assessed by the Visual Analog Scale (VAS) | Weekly from 1-week post-operative until 3 months; monthly from 4-12 months
  Will measure average knee pain over a given timeframe from 0 to 10 cm visual analogue scale where 0 cm equals no pain and 10 cm indicates the most severe pain the patient could imagine. Higher numbers equal greater levels of reported pain.
Time to return to full duty | 12 months post-operative
  Measured by the time from post-operative timepoint to time of full clearance for military tasks
Difference between the Tindeq Progessor and CSMi HUMAC NORM in measuring peak isometric knee extensor torque. | At either month 3, 6, 9, or 12, Tindeq testing will occur 24-72 hours after the bilateral strength assessment using the CSMi HUMAC NORM.
  Peak isometric extensor torque (nm/kg).
Difference between the Tindeq Progessor and CSMi HUMAC NORM in measuring knee extensor rate of torque development. | At either month 3, 6, 9, or 12, Tindeq testing will occur 24-72 hours after the bilateral strength assessment using the CSMi HUMAC NORM.
  Rate of torque development (nm/s)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn M Gee, MD, Principal Investigator — Keller Army Community Hospital
Locations (1):
- Keller Army Community Hospital, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication
Access Criteria: request can be made to study contacts and will be reviewed by the study principal investigator and human research protections office.

REFERENCES:
- [Background] Guerra ON, Coyle TE. Dentistry and the Ellis Fischel State Cancer Hospital. J Mo Dent Assoc. 1978 Jun-Jul;58(6):54-9. No abstract available. PMID 280702
- [Background] Nemcok JC. An analysis of 353 vaginal deliveries: natural versus anesthesia. J Am Osteopath Assoc. 1980 Dec;80(4):247-53. No abstract available. PMID 7239962
- [Background] Hixon JE, Pijanowski GJ, Weston PG, Shanks RD, Wagner WC. Evidence for an oscillator other than luteinizing hormone controlling the secretion of progesterone in cattle. Biol Reprod. 1983 Dec;29(5):1155-62. doi: 10.1095/biolreprod29.5.1155. PMID 6686068
- [Background] Matsushita N, Kato Y, Shimatsu A, Katakami H, Yanaihara N, Imura H. Effects of VIP, TRH, GABA and dopamine on prolactin release from superfused rat anterior pituitary cells. Life Sci. 1983 Mar 14;32(11):1263-9. doi: 10.1016/0024-3205(83)90196-0. PMID 6132313
- [Background] Marx RG, Stump TJ, Jones EC, Wickiewicz TL, Warren RF. Development and evaluation of an activity rating scale for disorders of the knee. Am J Sports Med. 2001 Mar-Apr;29(2):213-8. doi: 10.1177/03635465010290021601. PMID 11292048
- [Background] Herron P, Dykes R. The ventroposterior inferior nucleus in the thalamus of cats: a relay nucleus in the Pacinian pathway to somatosensory cortex. J Neurophysiol. 1986 Dec;56(6):1475-97. doi: 10.1152/jn.1986.56.6.1475. PMID 3806180
- [Background] Cobian DG, Koch CM, Amendola A, Williams GN. Knee Extensor Rate of Torque Development Before and After Arthroscopic Partial Meniscectomy, With Analysis of Neuromuscular Mechanisms. J Orthop Sports Phys Ther. 2017 Dec;47(12):945-956. doi: 10.2519/jospt.2017.7310. Epub 2017 Oct 9. PMID 28992769
- [Background] Pietrowa N, Jaczynowska Z, Duchowska H. [Treatment of uveitis in the course of rheumatoid arthritis in children]. Reumatologia. 1973;11(4):355-62. No abstract available. Polish. PMID 4768294
- [Background] Higgins LD, Taylor MK, Park D, Ghodadra N, Marchant M, Pietrobon R, Cook C; International Knee Documentation Committee. Reliability and validity of the International Knee Documentation Committee (IKDC) Subjective Knee Form. Joint Bone Spine. 2007 Dec;74(6):594-9. doi: 10.1016/j.jbspin.2007.01.036. Epub 2007 Aug 6. PMID 17888709
- [Background] Hill OT, Bulathsinhala L, Scofield DE, Haley TF, Bernasek TL. Risk factors for soft tissue knee injuries in active duty U.S. Army soldiers, 2000-2005. Mil Med. 2013 Jun;178(6):676-82. doi: 10.7205/MILMED-D-13-00049. PMID 23756076
- [Background] Behrend EI, Craig AM, Wilson SM, Denhardt DT, Chambers AF. Expression of antisense osteopontin RNA in metastatic mouse fibroblasts is associated with reduced malignancy. Ann N Y Acad Sci. 1995 Apr 21;760:299-301. doi: 10.1111/j.1749-6632.1995.tb44640.x. No abstract available. PMID 7785904
- [Background] Aguero AD, Irrgang JJ, MacGregor AJ, Rothenberger SD, Hart JM, Fraser JJ. Sex, military occupation and rank are associated with risk of anterior cruciate ligament injury in tactical-athletes. BMJ Mil Health. 2023 Nov 22;169(6):535-541. doi: 10.1136/bmjmilitary-2021-002059. PMID 35165197
- [Background] Hauret KG, Jones BH, Bullock SH, Canham-Chervak M, Canada S. Musculoskeletal injuries description of an under-recognized injury problem among military personnel. Am J Prev Med. 2010 Jan;38(1 Suppl):S61-70. doi: 10.1016/j.amepre.2009.10.021. PMID 20117601
- [Background] Molloy JM, Pendergrass TL, Lee IE, Hauret KG, Chervak MC, Rhon DI. Musculoskeletal Injuries and United States Army Readiness. Part II: Management Challenges and Risk Mitigation Initiatives. Mil Med. 2020 Sep 18;185(9-10):e1472-e1480. doi: 10.1093/milmed/usaa028. PMID 32107561
- [Background] Levine M, McElroy K, Stakich V, Cicco J. Comparing conventional physical therapy rehabilitation with neuromuscular electrical stimulation after TKA. Orthopedics. 2013 Mar;36(3):e319-24. doi: 10.3928/01477447-20130222-20. PMID 23464951